CLINICAL TRIAL: NCT00869518
Title: Randomized, Double-Blinded Evaluation of Rifabutin Based Therapy for Eradication of Staphylococcus Aureus Carriage in HIV Infected Individuals With Prior Skin and Skin Structure Infections
Brief Title: Rifabutin Based Therapy for the Eradication of Staphylococcus Aureus Colonization in HIV Infected Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08033578
Record Dates: First submitted 2009-03-24; First posted 2009-03-26 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-04

CONDITIONS: Staphylococcus Aureus; HIV Infections
Keywords: Staphylococcus aureus; colonization; eradication; HIV; rifabutin
MeSH Terms: conditions — Staphylococcal Infections; HIV Infections | interventions — Rifabutin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifabutin (Active Comparator): Subjects will be assigned to 7 days of treatment with rifabutin plus trimethoprim-sulfamethoxazole
  Interventions: Drug: rifabutin plus trimethoprim sulfamethoxazole
- Placebo (Placebo Comparator): Subjects will be assigned to 7 days of treatment with placebo plus trimethoprim-sulfamethoxazole
  Interventions: Drug: placebo plus trimethoprim-sulfamethoxazole

INTERVENTIONS:
Drug: rifabutin plus trimethoprim sulfamethoxazole — rifabutin 300 mg PO daily or equivalent depending on concomitant medications plus trimethoprim-sulfamethoxazole 1 DS tab twice daily both for 7 days
  Arms: Rifabutin
Drug: placebo plus trimethoprim-sulfamethoxazole — placebo plus trimethoprim-sulfamethoxazole 1 DS tab twice daily both for 7 days
  Arms: Placebo

SUMMARY:
DESIGN: This single center, double-blinded, randomized phase II study is being conducted to assess the efficacy of a rifabutin based regimen to eliminate S. aureus colonization in HIV infected individuals. Individuals must have HIV infection and a skin and skin structure infection (SSSI) in the prior 6 months to be eligible for screening. Prior to enrollment, subjects will be cultured for evidence of S. aureus colonization. Individuals who are culture positive at ≥ one body site will be eligible for enrollment. Subjects who meet inclusion and exclusion criteria and consent to participate in the study will be randomized to seven days of rifabutin plus trimethoprim-sulfamethoxazole (TMP-SMX) or TMP-SMX alone. Following completion of treatment subjects will be screened seven days, 30 days, and 60 days post-treatment for colonization at multiple body-sites. Subjects will also be actively followed for evidence of SSSI.

SUBJECT PARTICIPATION DURATION: 12 weeks

SAMPLE SIZE: 88 total subjects

POPULATION: 200 HIV infected individuals who receive care at San Francisco General Hospital HIV clinic (Ward 86) with a history of SSSI in the prior 6 months will be screened for S. aureus colonization.

DESCRIPTION OF AGENT OR INTERVENTION: This is a double-blind trial comparing rifabutin plus TMP-SMX versus placebo plus TMP-SMX. Placebo will be administered at a dose of 300 mg p.o. daily or an equivalent dose depending on co-administration of other drugs that may adjust the serum level of rifabutin. TMP-SMX will be administered at a dose of trimethoprim 160 mg and sulfamethoxazole 800 mg p.o. twice daily or adjusted per CrCl. Study drug will be provided by the study and administered for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. HIV infection as reported by the subject's physician
3. Physician-reported SSSI within the prior 6 months.
4. S. aureus colonization at ≥ 1 body site as defined as a positive culture for S. aureus at minimum one of five cultures taken at pre-enrollment screening.
5. Subjects (or their legally acceptable representatives) must have signed an informed consent documentation indicating that they understand the purpose of and procedures required for the study, and are willing to participate in the study

Exclusion Criteria:

1. Female subjects who are pregnant or lactating.
2. Known or suspected hypersensitivity to rifabutin, a rifamycin class antimicrobial, TMP-SMX or another sulfa based medication.
3. Known or suspected condition or concurrent treatment that would be contraindicated by the prescribing of rifabutin or TMP-SMX.
4. Receipt of an anti-staphylococcal antimicrobial within 14 days prior to administration of study drug (TMP-SMX, clindamycin, any macrolide, any tetracycline, any rifamycin, any fluoroquinolone, vancomycin, linezolid, daptomycin, any penicillin, any carbapenem, or any cephalosporin).
5. Diagnosis of an active SSSI or other signs and symptoms of S. aureus infection at the time of study enrollment
6. Physician-reported diagnosis of active or untreated latent mycobacterial infection
7. CrCl < 30 ml/min as determined by the Cockcroft-Gault Method using a serum creatinine from a value obtained within the last 6 months.
8. No serum creatinine value available for the subject in the SFGH clinical laboratory system (LCR) within 6 months prior to enrollment.
9. Physician-reported diagnosis of end-stage liver disease
10. Physician-reported diagnosis of uveitis in the past or at time of enrollment
11. Concomitant use of medications with unknown pharmacokinetic interactions with rifabutin or contraindicated with rifabutin (unboosted indinavir, unboosted saquinavir, delavirdine, atovaquone, azithromycin, Bacillus of Calmette and Guerin [only if recent administration for bladder cancer treatment], dapsone, dasatinib, erlotininb, ethinyl estradiol, fluconazole, imatinab, itinotecan, itraconazole, ixabepilone, lapatinib, levonorgestrel, mestranol, nilotininb, norelgestromin, norethindrone, posaconazole, ranolazine, sirolimus, sunitinib, tacrolimus, temsirolimus, trimetrexate, voriconazole, warfarin)
12. Colonizing S. aureus isolate resistant to TMP-SMX
13. Colonizing S. aureus isolate resistant to rifampin (rifampin resistance will serve as a surrogate for rifabutin resistance at initial screening)
14. Subjects who are unlikely to be able to comply with the mandated study visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry F Chambers, MD, Principal Investigator — University of Califronia, San Francisco; Brian S Schwartz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Rifabutin: Subjects assigned to 7 days of treatment with rifabutin plus trimethoprim-sulfamethoxazole
  rifabutin plus trimethoprim sulfamethoxazole: rifabutin 300 mg PO daily or equivalent depending on concomitant medications plus trimethoprim-sulfamethoxazole 1 DS tab twice daily both for 7 days
- Placebo: Subjects assigned to 7 days of treatment with placebo plus trimethoprim-sulfamethoxazole
  placebo plus trimethoprim-sulfamethoxazole: placebo plus trimethoprim-sulfamethoxazole 1 DS tab twice daily both for 7 days
Period: Overall Study
Arm/Group | Rifabutin | Placebo
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifabutin | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] | 42.3 [25 to 49] | 43.5 [25 to 63] | 42.9 [25 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Eradication of S. Aureus Colonization
Description: Eradication was measured by performing cultures for S aureus at the nose, throat, and groin
Time Frame: 30 days following completion of treatment
Measure: Number; unit: participants
Arm/Group | Rifabutin | Placebo
Number analyzed (Participants) | 5 | 5
participants | 0 | 0

2. Secondary Outcome: Eradication of S. Aureus Colonization
Description: Eradication was measured by performing cultures for S aureus at the nose, throat, and groin
Time Frame: 7 days following completion of treatment
Measure: Number; unit: participants
Arm/Group | Rifabutin | Placebo
Number analyzed (Participants) | 6 | 5
participants | 3 | 1

3. Secondary Outcome: Eradication of S. Aureus Colonization
Description: Eradication was measured by performing cultures for S aureus at the nose, throat, and groin
Time Frame: 60 days following completion of treatment
Population: Participants were colonized at day 30 (i.e. S. Aureus not eradicated) and were not checked again for follow-up.
Arm/Group | Rifabutin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Recurrent Skin and Skin Structure Infections (SSTI)
Description: recurrent SSTI was by self-report and exam, followed until positive colonization
Time Frame: up to 30 days following completion of treatment
Population: participants were followed until colonization; therefore, no participants were followed past 30 days
Measure: Number; unit: participants
Arm/Group | Rifabutin | Placebo
Number analyzed (Participants) | 6 | 6
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days after treatment
Arm/Group | Rifabutin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifabutin (N=6) | Placebo (N=6)
Hypersensitivity reaction (Immune system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes